CLINICAL TRIAL: NCT00008814
Title: Functional Magnetic Resonance Imaging (fMRI) in Infants
Brief Title: Functional Magnetic Resonance Imaging in Infants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Other Study IDs: NCRR-M01RR00400-0680
Record Dates: First submitted 2001-01-16; First posted 2001-01-18 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Healthy; Infant, Newborn, Diseases
Keywords: Cognition; Infant Development; MRI, Functional
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other

SUMMARY:
The study proposes to evaluate cognitive development in infants four months or younger by functional MRI and event related potential recording. fMRI imaging will be obtained following an auditory stimulus inside the 4 tesla magnet at the Center for Magnetic Resonance Research and will be correlated with ERP response to the same stimulus.

ELIGIBILITY:
Male or female infants less than 4 months old

Ages: 1 Day to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Institute of Child Development, Saint Paul, Minnesota, United States